CLINICAL TRIAL: NCT02369575
Title: Identification of Novel Markers of Human Lung Disease
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Megan Ballinger, Research Asst Professor, Ohio State University
Other Study IDs: 2014H0367
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: novel biomarkers of lung disease — we will be identifying molecular, genetic, and cellular markers of lung disease

SUMMARY:
The purpose of this study is to investigate new therapies for advanced lung disease.

DETAILED DESCRIPTION:
This research study is being conducted to learn about the progression and cause of lung disease. By agreeing to be a part of this study, you will allow the lung tissue which would normally have been discarded after your procedure, to be used for research purposes to allow us to understand more about your condition which may potentially lead to novel treatments and therapeutics. For this study, the investigators will isolate specific cells from the lung tissue and measure cellular, molecular and genetic mechanisms responsible for regulating lung disease. No other type of research will be performed on these samples nor will the samples be given to other investigators for unrelated research.

ELIGIBILITY:
Inclusion Criteria:

* any one on lung transplant list

Exclusion Criteria:

* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on lung transplant waiting list
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-07 (Actual)

PRIMARY OUTCOMES:
The development of novel therapeutics for interstial lung disease | 10 years
  Our research on these human lung cells will provide critical data which will aid in the diagnosis and treatment of a variety of different lung diseases, which have no cure.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ballinger, Principal Investigator — Ohio State University
Locations (1):
- Davis Heart and Lung Research Institute, Columbus, Ohio, United States